CLINICAL TRIAL: NCT01401816
Title: Advanced Provision of Emergency Contraception: Utilizing Technology to Increase Prescription Fill Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Alpert 3442-3
Record Dates: First submitted 2011-06-21; First posted 2011-07-25 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2011-06

CONDITIONS: Sexually Active
Keywords: Adolescents; Sexually Active; Unprotected Sex; Emergency Contraception
MeSH Terms: conditions — Unsafe Sex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Subjects in this group will receive a prescription for emergency contraception and then text-messages (on Day 1, 3 and 5 after enrollment) to their personal cell phone with a reminder to fill their prescription.
  Interventions: Other: Text Message
- Control Group (No Intervention): Subjects in this group will receive a only a prescription for emergency contraception and no reminder text messages.

INTERVENTIONS:
Other: Text Message — Subjects will receive a text message on their personal cell phone on Days 1, 3 and 5 after enrollment reminding them to fill their prescription.
  Arms: Intervention Group

SUMMARY:
Eighty-five percent of the 750,000 teenage pregnancies per year in the United States are unintended (Guttmacher Institute). Approximately half of all teenage pregnancies end in the birth of a child; the remaining proportion end in either abortion (30%) or miscarriage (20%). It has been estimated that if Emergency Contraception (Plan B) was used after every contraception failure, it could prevent 50% of unintended pregnancies and 60-70% of abortions annually.

Previous studies have showed the effectiveness of emergency contraception decreases with time after intercourse; the sooner it is taken-even if it means a matter of hours-the more effective it is in preventing pregnancy. Based on previous studies, it is clear that relying on obtaining emergency contraception on the same day or even the day after unprotected intercourse is not guaranteed. For example, approximately 27% of pharmacies called by the adolescent mystery caller did not have the medication available the day of the call and almost all of the pharmacies not stocking the medication would take greater than 24 hours to obtain it through their ordering system.

Thus, the concept of advanced provision of emergency contraception has been proposed to assure that the medication can be taken as soon as possible. Although this practice is known to be safe and has not shown any association with increased sexual risk or behaviors, it is unclear how often/if adolescents will fill a prescription for a medication that is not needed at the time of a medical encounter.

The investigators propose a randomized pilot study (n=60) of a text-messaging intervention that aims to increase the rate at which prescriptions for emergency contraception are filled. Based on practice norms in the BMC Adolescent Center, sexually active female adolescents (ages 13-21) in both the control and intervention groups will be provided a prescription for emergency contraception. The intervention group, however, will receive follow-up text message on their phone reminding them to fill the prescription.

Boston Medical Center Health Plan will provide prescription fill data regarding the prescriptions written at the time of enrollment. Approximately 6 weeks after enrollment, all study participants will be contacted for a follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Sexually Active
* Boston Medical Center Health Plan Insurance
* Personal Cell Phone

Exclusion Criteria:

* Pregnant
* Currently using a long-acting form of contraception (IUD, Depo, Implanon)
* No personal cell phone
* Insurance other than Boston Medical Center Health Plan

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Prescription Fill Rates | 1 month
  The primary outcome is whether the advanced provision prescription for emergency contraception is filled or not. This will be measured through insurance claims data obtained from BMC Health Plan a month after enrollment. Furthermore, the time to fill the prescription from the time of enrollment can be examined.

SECONDARY OUTCOMES:
Sexual Activity | 6 weeks
  Each study participant will receive a follow-up telephone call to his or her personal cell phone six weeks after enrollment to complete a follow-up survey that will consist of questions related to sexual activity since enrollment.
Contraception Use | 6 weeks
  Each participant will receive a follow-up telephone survey and answer questions regarding their use of contraception (if any) and how often they utilized such methods since enrollment.
Risk of Pregnancy | 6 weeks
  Each study participant will receive a telephone survey and be asked if they have used emergency contraception (EC) since enrolling in the study or if they have taken a pregnancy test since enrolling.
Knowledge of Emergency Contraception | 6 weeks
  Each study participant will receive a follow-up telephone survey and answer questions on the time-frame and accessibility of emergency contraception.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States